CLINICAL TRIAL: NCT02453971
Title: German Title: Prävention Substanzbezogener Störungen Bei Studierenden
Brief Title: Trial to Evaluate the Effects of the German eCHECKUP TO GO in Students
Acronym: PsSt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esslingen University of Applied Sciences (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIA5-2513DSM213
Record Dates: First submitted 2015-05-07; First posted 2015-05-27 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-06

CONDITIONS: Alcohol Consumption
Keywords: alcohol consumption; binge drinking; web-based personalized feedback program; students
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eCHUG-D (Experimental): The eCHUG group is requested to conduct the German Version of eCHECKUP TO GO and to fill in their code on the last page of the program.
  Interventions: Other: German Version of eCHECKUP TO GO
- control (No Intervention): It is an assessment only condition.

INTERVENTIONS:
Other: German Version of eCHECKUP TO GO — It is an online prevention program targeting alcohol consumption.
  Arms: eCHUG-D

SUMMARY:
The purpose of this study is to evaluate the effects of the German eCHECKUP TO GO (eCHUG-D) in students. Compared to the control group subjects who conducted eCHUG-D should have less alcohol consumption and less alcohol associated problems after three and six months.

DETAILED DESCRIPTION:
The effectivity of the eCHUG-D will be checked through a prospective randomized-controlled web-study.

All students at the participating universities will be informed about the PsSt-study. They have to agree to the informed consent to take part in the study. A missing agreement leads to exclusion. All subjects get an individual random login-code for study participation. After random assignment (intervention (eCHUG-D) vs. control group) all subjects have to answer the same web-questionnaires about their alcohol consumption (see outcome variables). Subjects of the intervention group are then requested to conduct eCHUG-D and to fill in their login-code at the end of the program.

The 3-month and 6-month follow-ups contain similar questions about alcohol consumption and alcohol related consequences. On 6-month follow-up additional questions ask about the acceptance of eCHUG-D (intervention group) and the acceptance of the study in general (control condition).

Earlier studies showed the effectiveness of eCHUG in US college samples. The primary endpoint of the study ist the amount of alcohol consumed. We hypothesize that the eCHUG group will show significantly lower levels of alcohol intake than the control group

ELIGIBILITY:
Inclusion Criteria:

* any student

Exclusion Criteria:

* ongoing recuperation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1465 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quantity-Frequency Questions (Alcohol Consumption) | 3-month
  Quantity of standard drinks during the last month and frequency of binge drinking occasions during the last month.
Quantity-Frequency Questions (Alcohol Consumption) | 6-month
  Quantity of standard drinks during the last month and frequency of binge drinking occasions during the last month.

SECONDARY OUTCOMES:
Maximum Blood Alcohol Concentration (BAC) | 3-month
  Estimation of BAC using the Widmark formula for the occasion during the past month when somebody drank the most.
Maximum Blood Alcohol Concentration (BAC) | 6-month
  Estimation of BAC using the Widmark formula for the occasion during the past month when somebody drank the most.
Rutgers Alcohol Problem Index (RAPI) (18-Item Version) | 3-month
  The RAPI is a 18-item self-administered screening tool for assessing adolescent problem drinking. Categorical answering is requested for consequences of alcohol use (0 = None,1 = 1-2 times, 2 = 3-5 times, 3 = More than 5 times). The RAPI is scored on a scale of 0-54.
Rutgers Alcohol Problem Index (RAPI) (18-Item Version) | 6-month
  The RAPI is a 18-item self-administered screening tool for assessing adolescent problem drinking. Categorical answering is requested for consequences of alcohol use (0 = None,1 = 1-2 times, 2 = 3-5 times, 3 = More than 5 times). The RAPI is scored on a scale of 0-54.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Heidenreich, PhD, Principal Investigator — University of Applied Sciences Esslingen
Locations (1):
- University of Applied Sciences Esslingen, Esslingen am Neckar, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Sobell, L. C., & Sobell, M. B. (2004). Alcohol consumption measures. In National Institute on Alcohol Abuse and Alcoholism, Assessing alcohol problems: A guide for clinicians and researchers (pp. 75-100). Bethesda, MD: Author.
- [Background] White HR, Labouvie EW. Towards the assessment of adolescent problem drinking. J Stud Alcohol. 1989 Jan;50(1):30-7. doi: 10.15288/jsa.1989.50.30. PMID 2927120
- See also: Link to the original web-site of the eCHUG and its contact information. — http://www.echeckuptogo.com